CLINICAL TRIAL: NCT00344071
Title: Pilot Study of Inflammatory Breast Cancer in Egypt and Tunisia
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904284; 04-C-N284
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-09-23

CONDITIONS: Inflammatory Breast Cancer
Keywords: Clinical; Tissue; Photographs; Women; Case-Control
MeSH Terms: conditions — Inflammatory Breast Neoplasms

SUMMARY:
One form of breast cancer, known as inflammatory breast cancer (IBC), is characterized by diffuse erythema (redness) and edema (peau d'orange) of the breast. This type of cancer is aggressive and poorly understood. It is rare in the United States (about 4 percent of cases), but more common in Egypt and Tunisia (up to 23 percent of cases). Conducting a case-control study of IBC is complicated by several factors, including the lack of standardized criteria for IBC. In addition, collecting pre-chemotherapy tissue and blood samples from IBC patients is difficult because treatment begins immediately after diagnosis.

In this pilot study, the National Cancer Institute will collaborate with two major cancer centers and two hospitals (in Egypt and Tunisia) to determine the feasibility of a case-control study of IBC. The study will assess the number and characteristics of IBC cases, the feasibility of identifying cases at diagnosis, and the availability of control subjects; will collect frozen pre-treatment tumor tissue from five IBC cases to determine whether RNA isolation is possible; will obtain digital photographs of the breasts of IBC cases; and will demonstrate collaboration between the institutions and personnel involved in the study. The study will last for approximately one year.

Participating hospitals will identify IBC cases. Consenting patients will undergo a breast examination in which the examining surgeon will complete an Initial Examination Form (IEF). Digital photographs of the breasts (but not face) will be taken and linked to the study ID number. Tissue examination results will be entered into the IEF. For five selected cases, additional pre-treatment tumor tissue will be collected and frozen.

This pilot study will assess the availability of controls for a case-control study by investigating the number and type of admissions to the Ear, Nose, and Throat and Ophthalmology Departments at participating hospitals during 2000-2003, using computerized records.

DETAILED DESCRIPTION:
Breast cancer characterized by diffuse erythema and edema, or peau d'orange, of the breast (inflammatory breast cancer (IBC)) is rare, particularly aggressive, and poorly understood. The extent of redness and edema or peau d'orange, of the breast required for a diagnosis of IBC has not been standardized. According to the most recent American Joint Committee on Cancer (AJCC) definition of inflammatory breast cancer, the signs of redness and edema or peau d'orange, should cover the majority of the breast, and should have arisen quickly. Breast cancers with redness and edema or peau d'orange, account for approximately 4 percent of breast cancers in the United States, but up to 23 percent of breast cancers in Egypt and Tunisia.

The proposed pilot study will determine the feasibility of conducting a case-control study of inflammatory breast cancer in collaboration with the National Cancer Institute-Cairo, Egypt, and the Institut Salah Azaiz, Tunis, Tunisia, the major cancer centers in Egypt and Tunisia, and Cairo University Hospital and Charles Nicolle Hospital, affiliated general hospitals from which controls will be selected. Currently, neither case study hospital collects data on the number of inflammatory breast cancer cases meeting the AJCC definition which will be used for the proposed case-control study. In addition, the geographic distribution of IBC cases at the two study hospitals (knowledge of which is necessary for the selection of appropriate controls) is unknown.

The goals of the pilot study are to assess the feasibility of the following critical components of the case-control study: 1) identifying a sufficient number of IBC cases at the time of diagnosis in the two study hospitals; 2) selecting appropriate hospital-based control subjects; 3) collecting frozen pre-treatment tumor tissue; 4) obtaining digital photographs of the breasts of IBC cases; and 5) communicating and working collaboratively with the study hospitals and personnel in Egypt and Tunisia. To accomplish these objectives, IBC cases meeting the AJCC definition as well as cases meeting other definitions of IBC will be identified over a one-year period at each of the two study hospitals. Computerized records at the control hospital for the years 2000-2003 will be used to enumerate the number of female patients with non-chronic diseases (and their age and geographic distribution) in the Departments of Ophthalmology and Ear, Nose and Throat (ENT). Pre-treatment frozen tumor tissue and digital photographs of the breast will be collected from five IBC cases at each study site.

ELIGIBILITY:
* INCLUSION CRITERIA:

All patients with redness and edema or peau d'orange, of the breast who are seen at the National Cancer-Cairo, Egypt or the Institute Salah Azair in Tunis, Tunisia during the period June 1, 2004 to May 31, 2005 will be eligible for the pilot study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250
Dates: Start 2004-09-08; Primary Completion 2007-04-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Egypt (2):
  - Cairo University Hospital, Cairo
  - National Cancer Institute-Cairo, Cairo
- Tunisia (2):
  - Association Tunisienne de lutte contre le Cancer (ATCC, le conseil, Tunis
  - Charles Nicolle Hospital, Tunisia, Tunis

REFERENCES:
- [Background] Attia-Sobol J, Ferriere JP, Cure H, Kwiatkowski F, Achard JL, Verrelle P, Feillel V, De Latour M, Lafaye C, Deloche C, et al. Treatment results, survival and prognostic factors in 109 inflammatory breast cancers: univariate and multivariate analysis. Eur J Cancer. 1993;29A(8):1081-8. doi: 10.1016/s0959-8049(05)80292-8. PMID 8518016
- [Background] Classon M, Settleman J. Emerging concepts in tumor progression and therapy. Semin Cancer Biol. 2000 Dec;10(6):393-7. doi: 10.1006/scbi.2000.0338. No abstract available. PMID 11170861
- [Background] Helal T, Nassiri M, Khalifa A. Immunohistochemical markers of tumor prognosis in breast cancer in Egypt. Cancer Detect Prev. 1997;21(3):201-6. PMID 9167036